CLINICAL TRIAL: NCT06790693
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Inavolisib Plus a CDK4/6 Inhibitor and Letrozole Versus Placebo Plus a CDK4/6 Inhibitor and Letrozole in Patients With Endocrine-Sensitive PIK3CA-Mutated, Hormone Receptor-Positive, HER2-Negative Advanced Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Inavolisib Plus CDK4/6 Inhibitor and Letrozole vs Placebo + CDK4/6i and Letrozole in Participants With Endocrine-Sensitive PIK3CA-Mutated, Hormone Receptor-Positive, HER2-Negative Advanced Breast Cancer
Acronym: INAVO123
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO45654; 2024-516162-11-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inavolisib + Letrozole + CDK4/6i (Experimental): Participants will receive inavolisib, letrozole and CDK4/6i.
  Interventions: Drug: Inavolisib; Drug: CDK4/6i; Drug: Letrozole
- Placebo + Letrozole + CDK4/6i (Placebo Comparator): Participants will receive placebo, letrozole and CDK4/6i.
  Interventions: Drug: Placebo; Drug: CDK4/6i; Drug: Letrozole

INTERVENTIONS:
Drug: Inavolisib — Participants will receive oral inavolisib once daily (QD).
  Other Names: GDC-0077; Itovebi
  Arms: Inavolisib + Letrozole + CDK4/6i
Drug: Placebo — Participants will receive oral placebo QD.
  Arms: Placebo + Letrozole + CDK4/6i
Drug: CDK4/6i — Participants will receive oral palbociclib on Days 1-21 of each 28-day cycle.
Drug: Letrozole — Participants will receive oral letrozole QD.

SUMMARY:
This study will evaluate the efficacy and safety of the combination of inavolisib plus a cyclin-dependent kinase 4 and 6 inhibitor (CDK4/6i) and letrozole versus placebo plus a CDK4/6i and letrozole in the first-line setting in participants with endocrine-sensitive PIK3CA-mutated hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-), advanced breast cancer (ABC).

ELIGIBILITY:
Inclusion Criteria:

* Women or men with histologically or cytologically confirmed carcinoma of the breast
* Documented ER-positive and/or progesterone receptor-positive tumor according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines
* Documented HER2-negative tumor according to ASCO/CAP guidelines
* De-novo HR+ , HER2- ABC, or, alternatively, relapsed HR+ , HER2- ABC after at least 2 years of standard neoadjuvant/adjuvant endocrine therapy without disease progression during that treatment and disease-free interval of at least 1 year since the completion of that treatment
* Participants who have bilateral breast cancers which are both HR-positive and HER2-negative
* Confirmation of biomarker eligibility
* Consent to provide fresh or archival tumor tissue specimen
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within the time frame in which contraception is required
* Metaplastic breast cancer
* Any prior systemic therapy for locally advanced unresectable or metastatic breast cancer
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Any history of leptomeningeal disease or carcinomatous meningitis
* Known and untreated, or active CNS metastases. Participants with a history of treated CNS metastases are eligible
* Active inflammatory or infectious conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye
* Symptomatic active lung disease
* History of or active inflammatory bowel disease
* Any active bowel inflammation
* Prior hematopoietic stem cell or bone marrow transplantation
* Treatment with strong cytochrome P450 (CYP) 3A4 inhibitors or strong CYP3A4 inducers within 4 weeks or 5 drug-elimination half-lives, prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2032-05-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 7 years)

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization to death from any cause (up to 7 years)
Investigator-assessed Objective Response Rate (ORR) | Up to 7 years
Investigator-assessed Duration of Response (DOR) | From the first occurrence of a confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 7 years)
Investigator-assessed Clinical Benefit Rate (CBR) | Up to 7 years
Time to Confirmed Deterioration (TTCD) in Pain | From baseline until end of follow-up (up to 7 years)
TTCD in Physical Function | From baseline until end of follow-up (up to 7 years)
TTCD in Role Function | From baseline until end of follow-up (up to 7 years)
TTCD in Global Health Status | From baseline until end of follow-up (up to 7 years)
Percentage of Participants with Adverse Events | From baseline until end of follow-up (up to 7 years)
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference with Daily Function of Symptomatic Treatment Toxicities Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 7 years
Number of Participants Reporting Each Response Option for Treatment Side-effect Bother Single-item General Population, Question 5 (GP5) from the Functional Assessment of Cancer Therapy-General Questionnaire; (FACT-G) | Up to 7 years
Change from Baseline in Symptomatic Treatment Toxicities as Assessed Through use of the PRO-CTCAE | Baseline up to 7 years
Change from Baseline in Treatment Side-effect Bother as Assessed Through use of the FACT-G GP5 Item | Baseline up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (204):
- United States (39):
  - Disney Family Cancer Center, Burbank, California
  - Scripps Health, La Jolla, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Ellison Institute of Technology, Los Angeles, California
  - Palo Alto Medical Foundation Research Center, Palo Alto, California
  - Kaiser Permanente - San Marcos, San Marcos, California
  - Palo Alto Medical Foundation Research Center, San Mateo, California
  - Palo Alto Medical Foundation Research Center, Sunnyvale, California
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Moffitt Cancer Center-McKinley Campus, Tampa, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Cancer Care Specialists of Central Illinois, O'Fallon, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Velocity Clinical Research, Annapolis, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - HCA Midwest Health, Kansas City, Missouri
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Cancer Clinic - Westside;Investigation Drug Services Pharmacy, Portland, Oregon
  - West Cancer Center, Germantown, Tennessee
  - Community Clinical Trials, Kingwood, Texas
  - Swedish Cancer Institute - Edmonds Campus, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute - Issaquah, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (5):
  - Centro Oncologico Korben, Caba
  - Centro Médico Fleischer, Capital Federal
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Instituto de Oncologia de Rosario, Rosario
  - Centro Oncológico de Excelencia, San Juan
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
- Brazil (13):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Santa Rita de Cassia Vitoria, Vitória, Espírito Santo
  - Obras Sociais Irma Dulce - Osid, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Centro de Oncologia de Alfenas, Alfenas, Minas Gerais
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Vencer Oncoclínica - Centro de Pesquisa do Piauí, Teresina, Piauí
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
- Canada (11):
  - Arthur J.E. Child Comprehensive Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - Unité de Recherche Clinique du CISSS de Laurentides, Saint-Jérôme, Quebec
- China (20):
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Peking Union Medical College Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Sun yat-sen University Cancer Center, Guangzhou
  - Sun Yat-Sen University Cancer Center - Huangpu Campus, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangmen Central Hospital, Jiangmen
  - Shandong Cancer Hospital, Jinan
  - Jinhua municipal central hospital, Jinhua
  - Yunnan Cancer Hospital, Kunming
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Shantou Center Hospital, Shantou
  - Tianjin Cancer Hospital, Tianjin
  - Tianjin Cancer hospital Airport hospital, Tianjin
  - Xinjiang Medical University Cancer Hospital, Ürümqi
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - Shanxi Provincial People's Hospital, Xi'an
- France (10):
  - Centre Oscar Lambret, Lille
  - Centre Cancerologie Grand Montpellier, Montpellier
  - INSTITUT CURIE_SITE PARIS - Service d'Oncologie Médicale., Paris
  - Centre CARIO - HPCA, Plérin
  - Chu La Miletrie, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - HOPITAL RENE HUGUENIN- Institut Curie, Saint-Cloud
  - Institut Universitaire de Cancer de Toulouse Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (15):
  - St. Elisabeth Krankenhaus Köln GmbH, Cologne
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - InVO - Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - Universitätsklinikum Münster, Münster
  - Klinikum Ernst von Bergmann, Potsdam
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Caritas Klinik St. Theresia -Frauenklinik Brustzentrum, Saarbrücken
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm Am Michelsberg, Ulm
- Italy (17):
  - Az. Osp. G. Panico, Tricase (LE), Apulia
  - A.O. S. Anna e San Sebastiano, Caserta, Campania
  - A.O. Universitaria Federico II Di Napoli, Napoli, Campania
  - U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Humanitas Centro Catanese Di Oncologia, Misterbianco (CT), Sicily
  - Azienda Sanitaria dell'Alto Adige;U.O.C. Oncologia Medic, Bolzano, Trentino-Alto Adige
  - Ospedale Civile - Livorno, Livorno, Tuscany
  - University of Eastern Piedmont - Maggiore della Carità University Hospital, Novara, Umbria
  - A.O. Santa Maria Terni, Terni, Umbria
- Japan (3):
  - Chiba Cancer Center, Chiba
  - Hokkaido University Hospital, Hokkaido
  - The Cancer Inst. Hosp. of JFCR, Tokyo
- Mexico (8):
  - Instituto Nacional De Cancerologia, Distrito Federal, Mexico CITY (federal District)
  - Hospital General de Mexico, MexicoCiudad de México, Nuevo León
  - Hospital Zambrano Hellion TecSalud, Monterrey, Nuevo León
  - Centro de Investigacion y Tratamiento Integral del Cancer: CITI Cancer Oaxaca S.A de C.V., Ciudad de Huajuapan de León, Oaxaca
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Centro Estatal de Cancerologia de Chihuahua, Chihuahua City
  - Iem-Fucam, D.F.
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
- Poland (10):
  - Instytut "Centrum Zdrowia Matki Polki", ?ód?
  - Bialostockie Centrum Onkologii, Bialystok
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Szpital Miejski Specjalistyczny Narutowicza, Krakow
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Wielkopolskie Centrum Onkologii im. Marii Sk?odowskiej-Curie, Późna
  - MRUKMED Lekarz Beata Madej-Mruk i Partner Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
  - Dolno?l?skie Centrum Onkologii, Wroc?aw
- PanOncology Trials, San Juan, Puerto Rico
- South Africa (3):
  - Linksfield Oncology Inc., Johannesburg
  - Abraham Oncology, Richards Bay
  - Wits Clinical Research, Soweto
- South Korea (9):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Soon Chun Hyang University Cheonan Hospital, Dongnam-gu, Cheonan-si
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (15):
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Navarra, Pamplona/iruña, Navarre
  - Hospital de Basurto, Bilbao, Vizcaya
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - IOB Madrid Institute of Oncology Hospital Beata Maria Ana de Jesus;Unidad Central de Oncología Médica y de Investigación Oncológica, Madrid
  - Hospital General Univ. Gregorio Maranon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria;Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
- Taiwan (6):
  - Chia-Yi Christian Hospital, Chiayi City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Uni Hospital, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Abdurrahman Yurtarslan Onkoloji Training and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Ba?c?lar Medipol Mega Üniversite Hastanesi, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Mersin City Education and Research Hospital, Mersin
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool
  - Western General Hospital, Edinburgh
  - Princess Alexandra Hospital, Harlow
  - St Bartholomew's Hospital, London
  - Royal Free Hospital, London
  - Mount Vernon & Watford Hospital Trust, Northwood
  - Churchill Hospital - Oxford Cancer & Haematology Centre, Oxford
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing